CLINICAL TRIAL: NCT06537388
Title: Comparison of High Frequency Jet Ventilation and Conventional Positive Pressure Ventilation for Endobronchial Ultrasound Examinations
Brief Title: High Frequency Jet Ventilation Versus Conventional Positive Pressure Ventilation for EBUS
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024173
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Intermittent Positive-Pressure Ventilation; High-Frequency Jet Ventilation; Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EBUS_cohort: All patients who underwent EBUS between January 1st 2019 and december 31st 2019 or January 1st 2023 and december 31st 2023 at Erasme University Hospital
  Interventions: Procedure: Ventilation type

INTERVENTIONS:
Procedure: Ventilation type — Type of ventilation used during the EBUS procedure, either HFJV or IPPV

SUMMARY:
Endobronchial ultrasound (EBUS) is frequently used in pneumology for diagnostic procedures like mediastinal biopsies. This procedure is usually done under general anesthesia. Different methods of ventilation are used according to center and physician preferences. In this retrospective study, complications of 2 types of ventilation will be analyzed:

* High frequency jet ventilation (HFJV)
* Conventional intermittent positive pressure ventilation (IPPV) Descriptive statistics will be used to present the data. Both ventilation techniques will be compared after propensity score matching. For HFJV patients from 2019 will be analyzed and for IPPV patients from 2023, as the team changed its practice over time.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent EBUS at Erasme University Hospital using either HFJV or IPPV between january 1st 2019 and december 31st 2019 or january 1st 2023 and december 31st 2023.

Exclusion Criteria:

* Incomplete medical chart
* Patients who expressed an opposition to the use of their medical data
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent EBUS for any indication at Erasme University Hospital using either HFJV or IPPV between january 1st 2019 and december 31st 2019 or january 1st 2023 and december 31st 2023.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Hypoxia | 24 hours
  defined as an SpO2 < 90% for more than 1 min
Severe hypoxia | 24 hours
  defined as an SpO2 (oxygen saturation by pulse oximetry) < 85% for more than 1 min
Hemodynamic instability | 24 hours
  defined as a systolic arterial blood pressure < 90/60 mm Hg
Cardiac arrythmia | 24 hours
  Any cardiac rhythm other than sinus rhythm
Laryngospasm | 24 hours
  Any occurence of laryngospasm
ICU admission | 24 hours
  Necessity for admission to the intensive care unit (ICU)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad KT, Sehgal IS, Gupta N, Singh N, Agarwal R, Dhooria S. Endoscopic ultrasound (with an echobronchoscope)-guided fine-needle aspiration for diagnosis of a mediastinal lesion in a mechanically ventilated patient: A case report and systematic review of the literature. Indian J Crit Care Med. 2016 Oct;20(10):608-612. doi: 10.4103/0972-5229.192057. PMID 27829719
- [Background] Anwar M, Fritze R, Base E, Wasserscheid T, Wolfram N, Koinig H, Hackner K, Lambers C, Schweiger T, Errhalt P, Hoda MA. Infraglottic versus supraglottic jet-ventilation for endobronchial ultrasound-guided transbronchial needle aspiration: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):999-1007. doi: 10.1097/EJA.0000000000001220. PMID 32453167
- [Background] Poling HE, Wolfson B, Siker ES. A technique of ventilation during laryngoscopy and bronchoscopy. Br J Anaesth. 1975 Mar;47(3):382-4. doi: 10.1093/bja/47.3.382. PMID 1138745
- [Background] Klain M, Smith RB. High frequency percutaneous transtracheal jet ventilation. Crit Care Med. 1977 Nov-Dec;5(6):280-7. doi: 10.1097/00003246-197711000-00007. No abstract available. PMID 338247
- [Background] Hautmann H, Gamarra F, Henke M, Diehm S, Huber RM. High frequency jet ventilation in interventional fiberoptic bronchoscopy. Anesth Analg. 2000 Jun;90(6):1436-40. doi: 10.1097/00000539-200006000-00034. PMID 10825336